CLINICAL TRIAL: NCT03731650
Title: Non-grafted Maxillary Sinus Floor Elevation With Simultaneous Implant Placement Using Different Implant Lengths
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdulnasser, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aaali.cairo university
Record Dates: First submitted 2018-09-12; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Maxillary Sinus Lift

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active comparator (Experimental)
  Interventions: Procedure: maxillary sinus lift
- placebo (Experimental)
  Interventions: Procedure: maxillary sinus lift

INTERVENTIONS:
Procedure: maxillary sinus lift — non grafted maxillary sinus floor augmentation with simultaneous implant placement

SUMMARY:
twenty recruited patients indicated for sinus augmentation and simultaneous implant placement will be divided into two groups (10 in each of the groups).to evaluate & compare bone formation & implant stability after shneiderian membrane elevation and augmentation with graft less tenting technique with different implant lengths.

group one will receive 8mm implant lenght while group two will receive 10mm implants.

ELIGIBILITY:
Inclusion Criteria:

* patient with atrophic maxilla & pneumatized maxillary sinus with residual bone height at least 4mm of residual ridge
* both sexes

Exclusion Criteria:

* patients with systematic diseases that may affect normal healing
* sinus pathology
* heavy smokers more than 20 cigarettes per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
height of gained bone | 6 months post operative
  two cone beam CT will be done for the patients, one immediate post operative & the other 6 months post operative then the amount of gained bone will be assessed by superimposing the same section in the two cone beam CT.

SECONDARY OUTCOMES:
implant stability | will be measured intra operative after implant insertion and will be measured once more 6 months post operative after the first operation at the time of implant exposure
  measurement of the implant stability using OSSTELL device.